CLINICAL TRIAL: NCT04711915
Title: Fixed Order, Open-Label, Dose-Escalation Study of DMT in Humans
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2000027720
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — N,N-Dimethyltryptamine

STUDY DESIGN:
Intervention Model Description: Healthy individuals and patients with major depressive disorder will participate in this study. Subjects will receive 0.1 mg/kg and 0.3 mg/kg DMT in a fixed order across 2 test days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.1 mg/kg DMT (Active Comparator): 0.1 mg/kg DMT administered intravenously
  Interventions: Drug: 0.1 mg/kg Dimethyltryptamine (DMT)
- 0.3 mg/kg DMT (Active Comparator): 0.3 mg/kg DMT administered intravenously
  Interventions: Drug: 0.3 mg/kg Dimethyltryptamine (DMT)

INTERVENTIONS:
Drug: 0.1 mg/kg Dimethyltryptamine (DMT) — 0.1 mg/kg DMT
  Other Names: Low Dose DMT
  Arms: 0.1 mg/kg DMT
Drug: 0.3 mg/kg Dimethyltryptamine (DMT) — 0.3 mg/kg DMT
  Other Names: Moderate Dose DMT
  Arms: 0.3 mg/kg DMT

SUMMARY:
The goal of this fixed order, open-label, dose-escalation study is to investigate the safety and efficacy of specific doses of dimethyltryptamine (DMT) in humans.

DETAILED DESCRIPTION:
The results of this study will inform the doses to be used in a larger, double-blind, randomized, placebo-controlled, crossover study. Since the goal of the open label study is to inform the double-blind, randomized, placebo-controlled study, the investigators are citing the hypothesis of the latter solely for providing context. The investigators hypothesize that the administration of DMT will result in neuroplastic changes in healthy and depressed subjects. These changes in neuroplasticity will be indexed using electroencephalographic (EEG) measures and tasks. These neuronal changes may in parallel cause changes in mood measured both in healthy and depressed subjects, which will be captured using appropriate psychometric measures of mood.

ELIGIBILITY:
Healthy controls inclusion criteria:

* Medically healthy
* Psychiatrically healthy

Healthy controls exclusion criteria:

* Unstable medical conditions
* Psychiatric illness

Depression inclusion criteria:

* Medically healthy
* Diagnosis of major depressive disorder

Depression exclusion criteria:

-Unstable medical conditions

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Pressure | -60 and -30 minutes before DMT administration; 0, +5, +10, +15, +20, +30, +45, +60, and +120 minutes after DMT administration
  Systolic and diastolic blood pressure will be measured before and several times after the administration of DMT on each test day.
Change in Heart Rate | -60 and -30 minutes before DMT administration; 0, +5, +10, +15, +20, +30, +45, +60, and +120 minutes after DMT administration
  Heart rate will be measured before and several times after the administration of DMT on each test day.
Change in Psychedelic Effects | -60 minutes before DMT administration; 0, +30, and +60 minutes after DMT administration
  The modified Altered States of Consciousness Rating Scale (ASC) will be used to assess drug-induced altered states of consciousness before and several times after drug administration. This is a 23-item subjective rating scale that will be completed using a visual analog scale format. Questions are scored 0 to 100 each; higher numbers indicate greater psychedelic effects.
Change in Anxiety | -60 minutes before DMT administration; 0, +30, and +60 minutes after DMT administration
  Anxiety will be assessed using a visual analog scale that subjects will be asked to score from 0 (not at all) to 100 (worst ever) to capture the net anxiety produced by DMT. This will be collected before and several times after DMT administration.
Drug Reinforcing Effects | +120 minutes after DMT administration
  Subjects will be asked to answer questions such as (1) How likely are you to use this drug? and (2) How much are you willing to pay for this experience? using a visual analog scale.
Overall Tolerability assessed by the VAS | +120 minutes after DMT administration
  Overall tolerability will be assessed using a visual analog scale that subjects will be asked to score from 0 (well tolerated) to 100 (intolerable) to capture the net tolerability of DMT.

CONTACTS AND LOCATIONS:
Locations (1):
- Biological Studies Unit at the VA Connecticut Healthcare System, Yale School of Medicine, West Haven, Connecticut, United States